CLINICAL TRIAL: NCT05227573
Title: Oxygen Partial Pressure and Lung Function After Orthopedic Surgery
Brief Title: PaO2 and Lung Function After Orthopedic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Profesor, Consultant surgeon, Umeå University
Other Study IDs: 233
Record Dates: First submitted 2022-01-24; First posted 2022-02-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Complications; Orthopedic Disorder
MeSH Terms: conditions — Postoperative Complications; Musculoskeletal Diseases | interventions — Orthopedic Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthopedic surgery — Knee-, hip-, shoulder- and elbow surgery

SUMMARY:
Hypoxia and reduced oxygen partial pressure is commonly occurring after abdominal surgery. This study aims to investigate whether similar changes also occur after orthopedic surgery in the form of upper limb surgery.

Inclusion: 60 patients undergoing orthopedic surgery in the form o knee-, hip-, shoulder- or elbow surgery.

Exclusion: Dementia or cognitive impairment that makes it impossible to participate in studies.

Arterial blood gas and lung function are undertaken before surgery, the day after surgery and at follow-up.

DETAILED DESCRIPTION:
Postoperative hypoxia complicates 30% - 50% of abdominal surgeries. People at particular risk for postoperative pulmonary complications including severe hypoxia are those who undergo abdominal surgery, emergency surgery or have a respiratory failure due to chronic lung disease including obstructive sleep apnea. The cause of postoperative restrictive lung function and hypoxia is unknown. Previous studies report that PaO2 decreases by an average of 2 kPa after abdominal surgery, while PaCO2 is unchanged and vital capacity decreases by 35%. The effect of orthopedic surgery on oxygen and carbon dioxide partial pressure and lung function has previously not been investigated. This study aims to investigate possible changes in oxygen partial pressure and vital capacity after orthopedic surgery.

Design: Prospective cohort study

Inclusion: 60 patients undergoing orthopedic surgery in the form o knee-, hip-, shoulder- or elbow surgery..

Exclusion: Dementia or cognitive impairment that makes it impossible to participate in studies.

Method: Blood gas measurements and Lung function (Vital capacity and FEV1) The day before surgery, the day after surgery and at follow-up.

Power analysis: There is a need to investigate 34 patients if the mean (SD) difference is 1 (2) kPa. Due to drop-outs the investigators calculate a need to include 60 patients.

Primary outcome measures:

• PaO2 from atrial blood gas

Secondary outcomes

* Vital capacity
* PaCO2 from atrial blood gas
* Forced expiratory volume in one second (FEV1)

Other variables examined: age, sex, height, weight, type of surgery, type of anesthesia, smoking status, length of surgery and previous diseases

ELIGIBILITY:
Inclusion Criteria: Patients undergoing shoulder or elbow surgery -

Exclusion Criteria: Dementia or cognitive impairment that makes it impossible to participate in studies. Not willing to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing shoulder or elbow surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen partial pressure | 1 day
  Change in oxygen partial pressure after surgery

SECONDARY OUTCOMES:
Vital capacity | 1 day
  Change in vital capacity after surgery
Oxygen partial pressure | 1 month
  Change in oxygen partial pressure after surgery
Carbon dioxide partial pressure | 1 day
  Change in carbon dioxide partial pressure after surgery
Carbon dioxide partial pressure | 1 month
  Change in carbon dioxide partial pressure after surgery
Vital capacity | 1 month
  Change in vital capacity after surgery
Forced expiratory volume in one second | 1 day
  Change in Forced expiratory volume in one second after surgery
Forced expiratory volume in one second | 1 month
  Change in Forced expiratory volume in one second after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, Prof, Principal Investigator — Surgical and Perioperative Sciences, Surgery, Umeå University, Sweden
Locations (1):
- Dept of Surgery, University hospital, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No